CLINICAL TRIAL: NCT04124458
Title: A Comparison of Pain Control AND Quality of Life Improvement Between Occipital Nerve Block And Occipital Nerve Radiofrequency Ablation: A Double-Blind Single Center Prospective Study
Brief Title: Occipital Nerve RF Between Occipital Nerve Block And Occipital Nerve Radiofrequency Ablation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Allevio Pain Management Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16397-11:07:0126-08-2019
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Occipital Neuralgia; Headache
MeSH Terms: conditions — Headache | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: This is a randomized, double blind, single-center, clinical trial. Participants will be randomly allocated to P-RF or occipital block intervention groups in a 1:1 ratio using a computer-generated algorithm. The study will be conducted over a period of 6 months, during which patients will make 4 visits (screening, baseline visit (Day 0) and 3, 6 months follow up visits, with ±1-week window). The study will be conducted at the Allevio Pain Clinic, Toronto, Canada. Research Ethics approvals will be sought.
Who Masked: Participant, Care Provider
Masking Description: Once eligible, the Redcap will assign the patient to one of the study group. Patients and physician provider will be blinded in the proposed study. Study questionnaires will be completed every three months by patients through RedCap System. Provider physician (here Dr.Rahul Shivaji Pathak) is the person who will perform the procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed Radiofrequency Ablation (Active Comparator): In radiofrequency ablation arm, sensory brunch of occipital nerve will be burn with max allowable temperature: 42 degrees Celsius, real temperature: 41 degrees Celsius, power=65 volts, two cycles of 180 second.
  Interventions: Device: Radiofrequency ablation
- Bilateral Occipital Nerve Block (Active Comparator): In this arm all steps are the same as other arm, except the generator will not be on and patient will have pain relief by injecting numbing medications beside the sensory nerves.
  Interventions: Device: Radiofrequency ablation

INTERVENTIONS:
Device: Radiofrequency ablation — In radiofrequency ablation arm, sensory brunch of occipital nerve will be burn with max allowable temperature: 42 degrees Celsius, real temperature: 41 degrees Celsius, power=65 volts, two cycles of 180 second.

SUMMARY:
This is a randomized, double blind, single-center, clinical trial. The study will be conducted over a period of 6 months. The study will be conducted at the Allevio Pain Clinic, Toronto, Canada.

DETAILED DESCRIPTION:
During the first visit the investigator will assess potential subject's eligibility. Screening and recruitment, and randomization, and administer questionnaires will be performed by research coordinator. Study informed consent form (ICF) can be signed on the RF procedure day. If additional visits will be required to finalize the procedures related to the first visit they will be scheduled accordingly. After randomization the qualified participants will be scheduled for their bilateral Occipital RF or bilateral Occipital Block.

Participants will be asked to complete the follow-up questionnaires at baseline, 3 and 6 months. On their last study visit, participants will have an exit interview, in addition to completing study measures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90
* Confirmed diagnosis of occipital headaches, patients with concurrent other types of headaches will not be excluded (except undiagnosed headaches)
* Duration of occipital headaches > 3 months

Exclusion Criteria:

* Non-English speakers;
* Refusal to sign informed consent;
* Allergy to medications which will be used in the study;
* Concurrent undiagnosed headaches
* Current brain tumors
* Current known tumors with known metastasis in other organs
* Occipital blocks within the last 3 months
* Currently receiving treatment with Botox for migraine.
* Patient has RF of occipital nerve/s within the last year

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-01-02 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life assessment: Short Form Brief Pain Inventory (BPI-SF) | Change from baseline BPI-SF at 6 months
  measured by Short Form Brief Pain Inventory (BPI-SF), between minimum of zero and maximum of ten

SECONDARY OUTCOMES:
At Least of 30% decrease in the pain score | Baseline, every 3 months up to 6 months
  measured by Visual Analog Scale (VAS), between minimum of zero and maximum of ten
At Least of 30% decrease in the pain score | Baseline, every 3 months up to 6 months
  measured by The Migraine Disability Assessment Test (MIDAS), between minimum of zero and maximum of twenty one
Quality of life assessment | Baseline, every 3 months up to 6 months
  measured by Beck's Depression Inventory (BDI)
Quality of life assessment: General Anxiety Disorder Questionnaire (GAD) | Baseline, every 3 months up to 6 months
  measured by General Anxiety Disorder Questionnaire (GAD)
Quality of life assessment: Patients self-reported perceived duration of effect (PSPDE) | Baseline, every 3 months up to 6 months
  measured by Patients self-reported perceived duration of effect (PSPDE)
Quality of life assessment: Global Improvement and Satisfaction score measured by PGIC) | Baseline, every 3 months up to 6 months
  measured by Global Improvement and Satisfaction score measured by PGIC)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 13. Cohen J. Statistical power analysis for the behavioral sciences. 2nd ed. Hillsdale, NJ: L. Erlbaum, 1988.
- [Result] Headache Classification Committee of the International Headache Society (IHS). The International Classification of Headache Disorders, 3rd edition (beta version). Cephalalgia. 2013 Jul;33(9):629-808. doi: 10.1177/0333102413485658. No abstract available. PMID 23771276
- [Result] Steiner TJ, Paemeleire K, Jensen R, Valade D, Savi L, Lainez MJ, Diener HC, Martelletti P, Couturier EG; European Headache Federation; Lifting The Burden: The Global Campaign to Reduce the Burden of Headache Worldwide; World Health Organization. European principles of management of common headache disorders in primary care. J Headache Pain. 2007 Oct;8 Suppl 1:S3-47. doi: 10.1007/s10194-007-0366-y. No abstract available. PMID 18034215
- [Result] Stovner Lj, Hagen K, Jensen R, Katsarava Z, Lipton R, Scher A, Steiner T, Zwart JA. The global burden of headache: a documentation of headache prevalence and disability worldwide. Cephalalgia. 2007 Mar;27(3):193-210. doi: 10.1111/j.1468-2982.2007.01288.x. PMID 17381554
- [Result] Ducic I, Felder JM 3rd, Fantus SA. A systematic review of peripheral nerve interventional treatments for chronic headaches. Ann Plast Surg. 2014 Apr;72(4):439-45. doi: 10.1097/SAP.0000000000000063. PMID 24374395
- [Result] Inan N, Inan LE, Coskun O, Tunc T, Ilhan M. Effectiveness of Greater Occipital Nerve Blocks in Migraine Prophylaxis. Noro Psikiyatr Ars. 2016 Mar;53(1):45-48. doi: 10.5152/npa.2015.10003. Epub 2016 Mar 1. PMID 28360765
- [Result] Okmen K, Dagistan Y, Dagistan E, Kaplan N, Cancan E. Efficacy of the greater occipital nerve block in recurrent migraine type headaches. Neurol Neurochir Pol. 2016;50(3):151-4. doi: 10.1016/j.pjnns.2016.01.015. Epub 2016 Feb 6. PMID 27154440
- [Result] Hascalovici JR, Robbins MS. Peripheral Nerve Blocks for the Treatment of Headache in Older Adults: A Retrospective Study. Headache. 2017 Jan;57(1):80-86. doi: 10.1111/head.12992. Epub 2016 Nov 30. PMID 27901275
- [Result] Kim DD, Sibai N. Prolongation of greater occipital neural blockade with 10% lidocaine neurolysis: a case series of a new technique. J Pain Res. 2016 Sep 29;9:721-725. doi: 10.2147/JPR.S112947. eCollection 2016. PMID 27729811
- [Result] Cohen SP, Peterlin BL, Fulton L, Neely ET, Kurihara C, Gupta A, Mali J, Fu DC, Jacobs MB, Plunkett AR, Verdun AJ, Stojanovic MP, Hanling S, Constantinescu O, White RL, McLean BC, Pasquina PF, Zhao Z. Randomized, double-blind, comparative-effectiveness study comparing pulsed radiofrequency to steroid injections for occipital neuralgia or migraine with occipital nerve tenderness. Pain. 2015 Dec;156(12):2585-2594. doi: 10.1097/j.pain.0000000000000373. PMID 26447705
- [Result] 11. Cervicogenic headache in Headache and Migraine Biology and Management 2015, Pages 203-212. Cooper W, Masih A.
- [Result] Dworkin RH, Turk DC, Wyrwich KW, Beaton D, Cleeland CS, Farrar JT, Haythornthwaite JA, Jensen MP, Kerns RD, Ader DN, Brandenburg N, Burke LB, Cella D, Chandler J, Cowan P, Dimitrova R, Dionne R, Hertz S, Jadad AR, Katz NP, Kehlet H, Kramer LD, Manning DC, McCormick C, McDermott MP, McQuay HJ, Patel S, Porter L, Quessy S, Rappaport BA, Rauschkolb C, Revicki DA, Rothman M, Schmader KE, Stacey BR, Stauffer JW, von Stein T, White RE, Witter J, Zavisic S. Interpreting the clinical importance of treatment outcomes in chronic pain clinical trials: IMMPACT recommendations. J Pain. 2008 Feb;9(2):105-21. doi: 10.1016/j.jpain.2007.09.005. Epub 2007 Dec 11. PMID 18055266